CLINICAL TRIAL: NCT00726375
Title: The Use of Etanercept (Enbrel) as Sole Treatment for Grade I Acute Graft Versus Host Disease
Brief Title: The Use of Etanercept Enbrel as Sole Treatment for Grade I Acute Graft Versus Host Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2007.139; HUM 17897 (Other: University of MI Medical School IRB)
Record Dates: First submitted 2008-07-28; First posted 2008-07-31 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-12

CONDITIONS: Acute Graft Versus Host Disease
Keywords: (GVHD)
MeSH Terms: conditions — Graft vs Host Disease | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etanercept (Experimental): a maximum of 8 SQ doses of 'Etanercept (Enbrel) at 0.4mg/kg per dose up to a maximum of 25 mg per dose
  Interventions: Drug: Etanercept (Enbrel)

INTERVENTIONS:
Drug: Etanercept (Enbrel) — Etanercept will begin within 72 hours of the diagnosis of Grade I acute GVHD and after consent for this study. Subjects receive eight doses of etanercept over four weeks. All doses will be administered by SQ injection. All subsequent doses will be given as subcutaneous injections into the skin. Injections will be given twice weekly with at least one day in between injections. The injections can be given in clinic, in the hospital, or self administered injections.

SUMMARY:
This is a clinical trial to see if treatment with etanercept for early skin graft-versus-host disease (GVHD) can effectively treat and prevent progression of the disease without using high dose steroids.

GVHD is a common complication following a bone marrow transplant from another donor. GVHD occurs after transplant, when the donor's blood cells (called lymphocytes) recognize parts of your body, such as the skin, as foreign. A certain chemical, called Tumor Necrosis Factor, or TNF, also causes damage to the skin. The main effect on the skin is a red rash, when the skin GVHD is mild, but in more severe forms the skin can blister.

We have been studying GVHD at the University of Michigan for the past decade. We know that high levels of TNF makes GVHD worse. Our research has shown that adding an anti-TNF drug (called etanercept or Enbrel®) to the standard GVHD treatment of high dose steroids leads to improvement in the GVHD in twice as many patients compared to when steroids alone are used. It is now standard practice at the University of Michigan and many other centers to treat GVHD with both steroids and etanercept.

The management of early skin GVHD for most patients involves treatment with steroids, given both as a cream and by either the mouth (in pills) or IV. Early skin GVHD is also called grade I GVHD, which means the skin rash covers less than half of the body. Steroid treatment can be effective; however, it also causes many complications such as an increased risk of infection, weight gain, stomach ulcers, muscle weakness and bone damage, among many others. We have developed this study to test whether starting treatment with etanercept and steroid creams alone can treat the GVHD without requiring the use of high dose steroids. The goal is to avoid the complications that come with high dose oral or IV steroid treatment. The high dose steroid treatment would only begin if your GVHD got worse.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have undergone HCT (donor cells from any source) with either a myeloablative or nonmyeloablative preparative regimen.
2. Patient may be any age.
3. Patient must have biopsy-proven Grade I acute GVHD (Appendix A). Biopsy report does not have to be back from Pathology prior to enrollment. Patients whose biopsy for GVHD identifies pathology inconsistent with GVHD will be removed from the study and replaced. However, because GVHD is a clinical diagnosis, biopsies which are non-diagnostic or do not show a clear non-GVHD etiology will not be cause to remove the patient from the study.

Exclusion Criteria:

1. Patients who are pregnant (positive urine or serum test) or nursing.
2. Active infections which are unresponsive to antibiotics (> 2 consecutive [at least 24 hours apart], positive blood cultures after initiation of treatment).
3. Allergic or otherwise undesirable reaction to etanercept.
4. Use of any oral or intravenous steroids at any previous time for GVHD treatment. Prior use of steroid therapy (i.e. hydrocortisone) as pre-medication for transfusions is permissible. Prior use of topical steroids is allowed.
5. Use of etanercept for any other purpose.
6. Noncompliance with medications.
7. Grade II-IV GVHD (history of or at time of study entry).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-05; Primary Completion 2013-07 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Choi, MD, Principal Investigator — The University of Michigan Comprehensive Cancer Center
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Gatza E, Braun T, Levine JE, Ferrara JL, Zhao S, Wang T, Chang L, Harris A, Pawarode A, Kitko C, Magenau JM, Yanik GA, Couriel DR, Goldstein S, Connelly J, Reddy P, Paczesny S, Choi SW. Etanercept plus topical corticosteroids as initial therapy for grade one acute graft-versus-host disease after allogeneic hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2014 Sep;20(9):1426-34. doi: 10.1016/j.bbmt.2014.05.023. Epub 2014 Jun 2. PMID 24892263

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Etanercept
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 51 [10 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 26
Race/Ethnicity, Customized [Number; unit: participants]
  White | 30
  Black or African American | 0
  Other | 4
Diagnosis [Number; unit: participants] — Cancer diagnosis.
  participants
    Acute myelogenous leukemia | 13
    Acute lymphoblastic leukemia | 6
    Multiple myeloma | 4
    Myelodysplastic syndrome | 4
    Non-Hodgkin's lymphoma | 2
    Myelofibrosis | 2
    Chronic lymphocytic leukemia | 1
    Chronic myelogenous leukemia | 0
    Nonmalignant disease | 2
Disease Risk Status [Number; unit: participants]
  Low | 13
  Intermediate | 5
  High | 16
Donor [Number; unit: participants]
  Matched related | 12
  Matched unrelated | 16
  Mismatched related | 0
  Mismatched unrelated | 6
CMV Status [Number; unit: participants] — Cytomegalovirus (CMV) status at baseline. R represents recipient status and D represents donor status.
  participants
    R+, D+ | 9
    R+, D- | 12
    R-, D+ | 3
    Recipient and donor negative | 10

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Who Progress Within 28 Days of Initiation of Etanercept Treatment
Description: We hypothesized that treatment of grade 1 acute GVHD (Graft Versus Host Disease) with etanercept would reduce the proportion of patients who progressed to grade 2 to 4 acute GVHD within 4 weeks of diagnosis from 58%, historically observed at our institution, to 38%.
Time Frame: 28 days
Measure: Number; unit: percentage of patients
Arm/Group | Etanercept
Number analyzed (Participants) | 34
percentage of patients | 29

2. Secondary Outcome: The Number of Patients in Complete Remission (CR) at Four Weeks.
Description: Estimate the proportion of patients in complete remission (CR) at four weeks who remain alive and never require additional therapy four weeks after the last dose of etanercept.
  Complete remission is defined as the resolution of all manifestations of GVHD (Graft Versus Host Disease) within the first four weeks of treatment. All organs must have a Grade 0.
Time Frame: 28 days
Measure: Number; unit: patients
Arm/Group | Etanercept
Number analyzed (Participants) | 34
patients | 14

ADVERSE EVENTS:
Time Frame: Patients were followed for adverse events from the first day treatment until 14 days after the treatment was stopped.
Description: Patients typically develop numerous complications such as infections, chemotherapy and medication side effects as part of a typical bone marrow transplant. Therefore AEs and SAES that coincide with a typical transplant course, unless fatal, or possibly related to the investigational therapy, were not reported.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 3/34
Other Adverse Events (participants affected / at risk) | 3/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=34)
Fever Without Neutropenia (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Creatinine Elevated (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=34)
Hypertension (Cardiac disorders) | 1 (1)
Fever Without Neutropenia (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Bladder Infection (Renal and urinary disorders) | 1 (1)
Creatinine Elevated (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to difficulties obtaining approval for insurance coverage of the study drug, only 34 of 50 patients were enrolled. The study was terminated prematurely and findings were reported for 34 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes